CLINICAL TRIAL: NCT02719457
Title: the Relationship Between Spot Marching Exercise Test and Six Minute Walk Test in Patient With Chronic Obstructive Pulmonary Disease
Brief Title: Spot Marching Exercise Test in Chronic Obstructive Pulmonary Disease
Acronym: SMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Vatcharaporn Khaweephab, Khon Kaen Hospital, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HE581308
Record Dates: First submitted 2016-02-06; First posted 2016-03-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Exercise testing; COPD; Upper and Lower limb exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 minute walk test (6 MWT) (Other): patients will be perform the six minute walk test (6 mwt) to evaluate their exercise capacity.
  Interventions: Other: 6 minute walk test (6 MWT)
- spot marching test (SMT) (Other): patients will be perform the spot marching test (SMT) to evaluate their exercise capacity.
  Interventions: Other: Spot marching test (SMT)

INTERVENTIONS:
Other: 6 minute walk test (6 MWT) — 6 minute walk test is the standard testing for COPD patients to evaluate their exercise capacity
  Arms: 6 minute walk test (6 MWT)
Other: Spot marching test (SMT) — Spot marching test is a new test that developed to evaluate their exercise capacity of COPD patients. This test is alternative method and practical to evaluate exercise capacity. The main benefit of this testing is use a small area to test and movement pattern involve both arm and leg. We expect that SMT may make COPD patient to more dyspnea in a short period of exercise.
  Arms: spot marching test (SMT)

SUMMARY:
the aim of this study to assess the relationship and compare physiological response between spot marching exercise test and 6 minute walk test in patient with chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is caused by airway inflammation (increase airway resistance) and destroyed of alveoli (decrease elastic recoil) leading to air trapping (GOLD, 2013). Dyspnea is the most symptom of COPD, a consequence of air trapping. Furthermore, inflammation of COPD has not only been assessed in the airways and lung compartment, but also in the systemic circulation that so called "systemic effects of COPD" such as skeletal muscle atrophy and dysfunction and cardiovascular disease (Wouter, 2002). The occurrence of dyspnea and systemic effects of COPD result in activity and exercise limitation when disease progressive downward.

Exercise testing is the most common determination of exercise limitation and responsiveness of intervention in COPD. It has several exercise protocols including laboratory test and field test. Both test aim to investigate exercise capacity but laboratory test have more parameter detail than field test. In 2013 Borel et al, classified the exercise protocols into three categories by using the workload characteristic (incremental or constant) and the self-paced test. Self-paced test was developed to solve the disadvantage of Incremental and Constant work rate (laboratory test). Moreover,it reflect functional activity and is easy to use. Self-paced test that most famous test such as six minute walk test, step test and stepper test Six minute walk test (6-MWT) assesses distance walked as far as possible within 6 minutes on straight courses. Although the 6-MWT is the most reliable, but it is impractical (Kocks et al., 2011) because of environmental constrain (this test should be performed wild area).

Step test was performed in small area such as hospitals and physician's office. However, these protocols have a risk of falling. Therefore, it was unsuitable for patients who have the imbalance or articular problem.

In 2010, Borel et al., developed six-minute stepper test (6-MST) to solve problem of 6MWT and step test. This study reported that 6-MST used oxygen consumption (VO2) lower than 6MWT. They reasoned that during stepper test, subject move upper limb fewer than walking test. Similarly with Mayo et al., 2001, they found heart rate and expiratory minute ventilation (VE) response of arm performance higher than leg. Therefore, movement of the upper limbs may be increase VO2 peak during exercise test of COPD patient.

Exercise limitation in COPD patient is not only occurs in lower body activity but also occurs during upper task due to systemic effect of disease. Upper body activity was used in daily activity such as lifting, bathing and washing. The almost protocols of exercise test were focused on lower limb test.

The investigators need to find the exercise tests which have the performance in both of upper and lower part movement and are easy to apply in a small setting. In 2013, Premsri et al. studied marching exercise on sympathetic activation in sedentary Thais. And in 2013, Promsrisuk et al. study effects of brisk marching on anthropometry, functional exercise capacity and physical performance among elderly women. Marching exercise have repetitive pattern of arm and leg alternated movement by bending hip between 45-90 degree with knee flexion (Premsri et al.,2013) and also lifting their shoulder flexion up at 90 degree.

Therefore, The investigators interested in the pattern of marching exercise that use both upper and lower extremity and used for exercise test in COPD patient. The investigators expect that marching can increase the performance at maximum level nearby 6-MWT COPD is a major disease in Thailand that not only affects the quality of life for the patient but also is a burden for their family and society at large in terms of the costs of health care and loss of economic activity. Improvements in diagnosis care and treatment can help to minimize the problems but the first stage is diagnosis and assessment. Despite the fact that there are many different exercise protocols that have been used for this purpose there is still an need for a test that is easy to use, especially in the community, and one that involves both arms and legs and is more representative of the activity of daily life. This project is concerned with developing such a test.

Therefore, this study to assess the relationship and compare physiological response between spot marching exercise test and 6 minute walk test in patient with chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* mild to very severe COPD patients

Exclusion Criteria:

* Exacerbate within a month prior, which was a cause of admission to the hospital emergency room or been admitted to hospital.
* Are changed medicines within a month ago.
* Have been used home oxygen therapy.
* Have musculoskeletal or neuromuscular problem affecting balance and walking.
* Using walking aid device.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
number of step of Spot Marching Test | up to 6 min

SECONDARY OUTCOMES:
Heart rate | every minute at pre-exercise for 5 min, during exercise test for 6 min and recovery phase for 10 min
Electrocardiogram (lead II) | every minute at pre-exercise for 5 min, during exercise test for 6 min and recovery phase for 10 min
Respiratory rate | every minute at pre-exercise for 5 min, during exercise test for 6 min and recovery phase for 10 min
Blood pressure | up to 2 minute in recovery phase
  include , systolic blood pressure, diastolic blood pressure, mean arterial pressure
peripheral oxygen saturation (SpO2) | every minute at pre-exercise for 5 min, during exercise test for 6 min and recovery phase for 10 min
partial pressure of end tidal carbondioxide | every minute at pre-exercise for 5 min, during exercise test for 6 min and recovery phase for 10 min
number of step of 6 minute walk test | up to 6 min
distance of 6 minute walk test | up to 6 min

CONTACTS AND LOCATIONS:
Overall Officials: Vatcharaporn Khaweephab, Master, Principal Investigator — school of physical therapy,faculty of associated medical sciences
Locations (2):
- Thailand (2):
  - Khon Kaen Hospital, Khon Kaen, Changwat Khon Kaen
  - Khonkaen univercity, Khonkaen, Khonkaen